CLINICAL TRIAL: NCT03368196
Title: Phase 1, Multicenter, Open-label Study of DS-8201a to Assess Safety and Pharmacokinetics in Subjects With HER2-Positive Advanced and/or Refractory Gastric, Gastroesophageal Junction Adenocarcinoma, or Breast Cancer
Brief Title: DS-8201a in Patients With Cancer That Tests Positive for Human Epidermal Growth Factor Receptor 2 (HER2) Protein
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Taiwan Ltd., a Daiichi Sankyo Company (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-A-A103
Record Dates: First submitted 2017-12-04; First posted 2017-12-11 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Adenocarcinoma, Gastric; Neoplasm, Breast
Keywords: Stomach cancer; Cancer where the esophagus meets the stomach; Human epidermal growth factor 2; HER2; Breast Cancer; Adenocarcinoma, Gastroesophageal Junction (GEJ); Gastric Cancer; Antibody drug conjugate (ADC); Oncology
MeSH Terms: conditions — Adenocarcinoma; Breast Neoplasms; Stomach Neoplasms; Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DS-8201a (Experimental): DS-8201a administered by intravenous infusion on Day 1 of each cycle, once every 3 weeks (Q3W)
  Interventions: Drug: DS-8201a

INTERVENTIONS:
Drug: DS-8201a — An antibody drug conjugate

SUMMARY:
HER2-positive cancer is a cancer that tests positive for a protein called human epidermal growth factor receptor 2 (HER2). HER2 promotes the growth of certain cancer cells. This study will test DS-8201a (trastuzumab deruxtecan), a HER2-targeted antibody and topoisomerase I inhibitor conjugate.

The safety and tolerability profile of DS-8201a will be assessed in Chinese patients with certain types of stomach and breast cancer that test positive for HER2. It also will test how DS-8201a moves within the body (pharmacokinetics).

DETAILED DESCRIPTION:
The expected time from the first subject's enrollment until the last subject's enrollment is approximately 8 months. The screening period is 28 days and each cycle of treatment is 21 days.

The number of treatment cycles is not fixed in this study. Subjects who continue to derive clinical benefit from the study drug in the absence of withdrawal of consent, progressive disease (PD), or unacceptable toxicity may continue the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Has a pathologically documented unresectable or metastatic gastric or GEJ adenocarcinoma, or breast cancer, with HER2 expression [immunohistochemistry (IHC) 3+, 2+, or 1+ and/or in situ hybridization (ISH) +] that is refractory to or intolerable with standard treatment, or for which no standard treatment is available
* Has a left ventricular ejection fraction (LVEF) ≥ 50%
* Has an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1

Exclusion Criteria:

* Has a medical history of myocardial infarction within 6 months before enrollment
* Has a medical history of ventricular arrhythmias, other than rare occasional premature ventricular contractions
* Has uncontrolled or significant cardiovascular disease
* Has any other history or condition that might compromise:

  1. Safety of the participant or offspring
  2. Safety of study staff
  3. Analysis of Results

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 participants who met all inclusion criteria and no exclusion criteria were enrolled and received treatment in Taiwan.
Pre-assignment Details: The 6.4 mg/kg DS-8201a dose was chosen for this study based on the efficacy, safety, and pharmacokinetic profiles established in an earlier Phase 1 trial.
Groups:
- DS-8201a: Participants who received 6.4 mg/kg DS-8201a administered by intravenous infusion on Day 1 of each cycle, once every 3 weeks.
Period: Overall Study
Arm/Group | DS-8201a
Started | 12
Completed (Ongoing as of data cutoff 14 Sept 2018) | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline demographics were assessed in the Safety Analysis Set.
Arm/Group | DS-8201a
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 12

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events Following Treatment With DS-8201a (Trastuzumab Deruxtecan)
Description: Adverse events (AEs) were to be coded using MedDRA Version 20.1 and assigned severity grades based on Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. A treatment-emergent adverse event (TEAE) was defined as an AE that occurred, having been absent before the first dose of study drug, or had worsened in severity or seriousness after initiating the study drug until 47 days after last dose of study drug.
Time Frame: Baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever came first), up to approximately 5 months post-dose
Population: Treatment-emergent adverse events (TEAEs) were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a
Number analyzed (Participants) | 12
Participants
  Any TEAE | 12
  Any drug-related TEAE | 12
  Any TEAE of CTCAE Grade ≥3 | 7
  Any drug-related TEAE of CTCAE Grade ≥3 | 6
  Any serious TEAE | 2
  Any drug-related serious TEAE | 1
  Any serious TEAE of CTCAE Grade ≥3 | 2
  Any drug-related serious TEAE of CTCAE Grade ≥3 | 1
  Any TEAE leading to drug withdrawal | 0
  Any TEAE leading to dose reduction | 2
  Any drug-related TEAE leading to dose reduction | 2
  Any TEAE leading to dose interruption | 5
  Any drug-related TEAE leading to dose interruption | 5
  Any TEAE leading to death | 0

2. Secondary Outcome: Pharmacokinetic Parameter of Maximum (Peak) Observed Serum Concentration (Cmax) Following Cycle 1 and Cycle 3 Treatment With DS-8201a (Trastuzumab Deruxtecan)
Description: Maximum concentration (Cmax) of DS-8201a and total anti-HER2 antibody was assessed.
Time Frame: Cycles 1 and 3, Day 1: before infusion (BI), end of infusion (EOI), 2 hours, 4 hours, 7 hours; Days 2 and 4, 24 hours, 72 hours; Days 8, and 15; Cycles 2, 4, 6 and 8, Day 1: BI and EOI
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | DS-8201a
Number analyzed (Participants) | 12
ug/mL
  DS-8201a, Cycle 1 | 157 (19.1)
  DS-8201a, Cycle 3: number analyzed (Participants) | 10
  DS-8201a, Cycle 3 | 163 (19.5)
  Total Anti-HER2 antibody, Cycle 1 | 150 (22.6)
  Total Anti-HER2 antibody, Cycle 3: number analyzed (Participants) | 10
  Total Anti-HER2 antibody, Cycle 3 | 154 (16.6)

3. Secondary Outcome: Pharmacokinetic Parameter of Maximum (Peak) Observed Serum Concentration (Cmax) of MAAA-1181a Following Cycle 1 and Cycle 3 Treatment With DS-8201a (Trastuzumab Deruxtecan)
Description: Maximum concentration (Cmax) of MAAA-1181a was assessed.
Time Frame: as for outcome 2
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DS-8201a
Number analyzed (Participants) | 12
ng/mL
  MAAA-1181a, Cycle 1 | 11.9 (3.79)
  MAAA-1181a, Cycle 3: number analyzed (Participants) | 10
  MAAA-1181a, Cycle 3 | 9.01 (1.36)

4. Secondary Outcome: Pharmacokinetic Parameter of Area Under the Serum Concentration-time Curve During Dosing Interval (AUCtau) Following Cycle 1 and Cycle 3 Treatment With DS-8201a (Trastuzumab Deruxtecan)
Description: Area under the serum concentration-time curve during dosing interval (AUCtau) of DS-8201a and total anti-HER2 antibody was assessed.
Time Frame: as for outcome 2
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug*d/mL
Arm/Group | DS-8201a
Number analyzed (Participants) | 12
ug*d/mL
  DS-8201a, Cycle 1 | 631 (173)
  DS-8201a, Cycle 3: number analyzed (Participants) | 10
  DS-8201a, Cycle 3 | 991 (109)
  Total Anti-HER2 antibody, Cycle 1 | 821 (312)
  Total Anti-HER2 antibody, Cycle 3: number analyzed (Participants) | 10
  Total Anti-HER2 antibody, Cycle 3 | 1180 (208)

5. Secondary Outcome: Pharmacokinetic Parameter of Area Under the Serum Concentration-time Curve During Dosing Interval (AUCtau) of MAAA-1181a Following Cycle 1 and Cycle 3 Treatment With DS-8201a (Trastuzumab Deruxtecan)
Description: Area under the serum concentration-time curve during dosing interval (AUCtau) of MAAA-1181a was assessed.
Time Frame: as for outcome 2
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*d/mL
Arm/Group | DS-8201a
Number analyzed (Participants) | 12
ng*d/mL
  MAAA-1181a, Cycle 1 | 36.1 (9.71)
  MAAA-1181a, Cycle 3: number analyzed (Participants) | 10
  MAAA-1181a, Cycle 3 | 41.3 (5.06)

6. Secondary Outcome: Best Overall Response By The Investigator's Assessment (Unconfirmed) in Participants With HER2-Positive Advanced and/or Refractory Gastric, Gastroesophageal Junction Adenocarcinoma, or Breast Cancer
Description: Best overall response (BOR) was assessed by the investigator based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. Complete response (CR) was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Time Frame: as for outcome 1
Population: Response was assessed in the Response Evaluable Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a
Number analyzed (Participants) | 11
Participants
  Complete response (CR) | 0
  Partial response (PR) | 4
  Stable disease (SD) | 7
  Non-Complete Response (CR)/Non-Progressive Disease (PD) | 0
  Progressive Disease (PD) | 0
  Non-evaluable (NE) | 0

7. Secondary Outcome: Objective Response Rate (Unconfirmed) As Assessed in Participants With HER2-Positive Advanced and/or Refractory Gastric, Gastroesophageal Junction Adenocarcinoma, or Breast Cancer
Description: Objective response rate (ORR; defined as participants who achieved CR and PR) was assessed by the investigator based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: as for outcome 1
Population: Response was evaluated in the Response Evaluable Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a
Number analyzed (Participants) | 11
Participants | 4

8. Secondary Outcome: Disease Control Rate (Unconfirmed) As Assessed in Participants With HER2-Positive Advanced and/or Refractory Gastric, Gastroesophageal Junction Adenocarcinoma, or Breast Cancer
Description: Disease control rate (DCR; defined as participants who achieved CR, PR, and SD) was assessed by the investigator based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: as for outcome 1
Population: Response was evaluated in the Response Evaluable Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-8201a
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from baseline up to withdrawal of consent, progressive disease, or unacceptable toxicity (whichever came first), up to approximately 5 months.
Arm/Group | DS-8201a
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-8201a (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DS-8201a (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Punctate keratitis (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 3
Influenza like illness (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Cellulitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Platelet count decreased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 6
White blood cell count decreased (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 3
Weight decreased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Ejection fraction decreased (Investigations) | 1
Liver function test increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/96/NCT03368196/Prot_SAP_001.pdf